CLINICAL TRIAL: NCT05580432
Title: The Effect of Parenting With Positive Behavior Interventions on Community Inclusion for Military Connected and Dependent Children With Autism and Their Parents
Brief Title: Effect of Parenting With Positive Interven on Comm Inclusion for Military Connected and Dependents With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20025356
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Waitlisted control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate behavioral intervention (Experimental): Participants will receive the intervention immediately
  Interventions: Behavioral: Parenting with Positive Behavior Interventions
- Delayed behavioral intervention (Active Comparator): Participant will receive the intervention after a 12 month delay
  Interventions: Behavioral: Parenting with Positive Behavior Interventions

INTERVENTIONS:
Behavioral: Parenting with Positive Behavior Interventions — Parenting with Positive Behavior Interventions is a 5 month packaged intervention. The curriculum and each element of the training and coaching program is described in detail below.
  Each month, participants will participate in the following five activities:
  1. Didactic Training: Participants will view a presentation
  2. Workbook/Homework: Participants will complete a guided worksheet
  3. Coaching Meeting - Planning: Participants will meet with a coach who is an expert in autism and behavior
  4. Coaching - Observation/ Feedback: The coach will observe parent implementing the strategy, then provide feedback and direction regarding use of technique
  5. Virtual Parent Community of Support Meeting: Attend parent led community support meeting to network, share experiences and information, and exchange ideas

SUMMARY:
The purpose of this research study is to find out if a training program for parents with military dependent or connected children with autism (ASD) who have challenging behavior will help those children and their families participate in more community activities. The training program, called Parenting with Positive Behavior Interventions, may help military parents learn new tools that will help their children with autism and challenging behavior attend community activities more easily.

DETAILED DESCRIPTION:
Participants will be randomly assigned (like the flip of a coin) to either immediately receive the Parenting with Positive Behavior Interventions or you will be asked to wait in a control condition for six months and then receive the same intervention. Participants have an equal chance of being assigned to any one of the groups (get the treatment immediately or wait 6 months) but will be given a chance to receive the intervention regardless within 6 months.

In this study, participants will be asked to do the following things:

1. Attend (virtually or in-person) a one-hour monthly training about behavior interventions for children with autism.
2. Participate in two 60- minutes sessions with a behavior coach (virtually or in-person) each month to talk about a community goal they want to complete with their child.
3. Attend an optional 60-minute meeting with other research participates each month to talk about their experience learning how to manage their child's behavior.
4. Work with a researcher to fill out a series of questionnaires 3 times during the study. These questionnaires will ask about participants, their child's challenging behaviors, stress related to community activities with their child, and how often they participate in community activities with their child with autism and challenging behavior.

ELIGIBILITY:
Inclusion Criteria:

Parent Inclusion Criteria:

1. Be older than 18 years
2. a. Serve or be the partner of a person who serves (or served, in the case of a deceased member) in the military(active duty, retired, medically discharged, deceased or on reserves) b. Be connected to the military (works as a civilian on base, works as a federal employee to provide services on base, provides services to the military, or is a contractor with the military OR has an immediate family member other than the parent who lives with the child and is active duty, retired, medically discharged, deceased or on reserves)
3. Be the parent of a child with ASD who is between the ages of 5 - 11
4. Be able to provide consent to participate

Child inclusion criteria:

1. Be a military dependent child (a military dependent child is a child with a parent, step-parent or guardian who is currently serving in, retired or medically discharged from the Army, Navy, Air Force, Marines, Coast Guard, or the National Guard on active duty or reserves or a parent or guardian died in service of one of the branches of military listed above.)
2. Be a military connected child (a child whose parent works as a civilian on base, works as a federal employee to provide services on base, provides services to the military, or is a contractor with the military OR a child who has an immediate family member other than the parent who lives with the child and is active duty, retired, medically discharged, deceased or on reserves)
3. Have a medically diagnosed and/or educational eligibility label of autism, autism spectrum disorder, or any other condition associated with autism
4. Display challenging behavior at home or in the community.
5. Be between the ages of 5 - 11

Exclusion Criteria:

Parent Exclusion Criteria:

1. Be unwilling or unable to consent to participate
2. Be unwilling or unable to provide consent for their child with ASD to participate
3. Be unwilling or unable to participate in the intervention

Child Exclusion Criteria:

1. Not living with the parent who is participating in the intervention
2. Hospitalized or in residential treatment outside of the parent's home

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Change in frequency of child with ASD's challenging behavior | Baseline to 12 months
  The Behavior Problems Inventory (BPI-01) records the frequency of a child with ASD's challenging behavior on a 4-point scale (never, monthly, weekly, daily). Responses for each item are summed to yield three subscale frequency scores, Self-Injurious Behavior, Stereotyped Behavior, and Aggressive/Destructive Behavior
Change in severity of child with ASD's challenging behavior | Baseline to 12 months
  The BPI-01 records the severity of a child with ASD's challenging behavior on a 3- point scale (Mild, Moderate, Severe). Item responses are summed to yield three subscale severity scores, Self-Injurious Behavior, Stereotyped Behavior, and Aggressive/Destructive Behavior

SECONDARY OUTCOMES:
Change in frequency of participation by child with ASD | Baseline to 12 months
  The Participation and Environment Measure - Children and Youth (PEM-CY) records the frequency of a child's frequency of participation in everyday activities. The survey asks about 25 types of activities. Parents rate how often the child has participated in the activity over the past 4 months on an 8-point scale (never to once in the last 4 months). Item responses are summed to yield three subscale frequency scores, home, school, and community.
Change in involvement during participation by child with ASD | Baseline to 12 months
  PEM-CY records the level of involvement during a child's participation in everyday activities. The survey asks level of involvement for 25 types of activities. Parents rate how involved the child was while participating in the activity over the past 4 months on an 5-point scale (very involved to minimally involved). Item responses are summed to yield three subscale involvement scores, home, school, and community.
Change in parent desire for change in participation by child with ASD | Baseline to 12 months
  PEM-CY records the degree to which a parent would like a child's participation in everyday activities to change. The survey asks about 25 types of activities. Parents check all changes desired (no change desired; yes, do more often; yes, do less often; yes, be more involved; yes, be less involved). Item responses are summed to yield three subscale involvement scores, home, school, and community.
Change in environmental support for participation by child with ASD | Baseline to 12 months
  PEM-CY records the situational resources that may help or hinder a child's participation in everyday activities. The survey asks about 45 different resources. Parents mark the degree to which resources are needed/helpful on a 4-scale. Item responses are summed to yield three subscale involvement scores, home, school, and community.
Change in community participation by parents | Baseline to 12 months
  The Participation in Meaningful Life Roles for Parents of Children with ASD records the degree to which parents of children with ASD are able to engage in life roles that are meaningful to them, such as working a job, volunteering, interacting with family members, engaging in community recreation, etc. Parents complete this measure using a 6 point likert scale.
Change in parental stress | Baseline to 12 months
  The Parental Stress Scale (PSS) measures parents feelings and perceptions about their relationship with their child using 17 questions. Parents rate each question from 1-strongly disagree to 5-strongly agree. Ratings are summed to yield a single score with higher numbers indicating more stress
Change in child's behavior | Baseline to 12 months
  Parents will rate their child's behavior using the age appropriate version of the Strengths and Difficulties Questionnaire (SDQ). The survey contains 25 to 27 behaviors which parents rate as no, a little, or a lot. Scores are summed to yield a single score.
Change in child's response to behavior | Baseline to 12 months
  Parents will rate their child's response to their own behavior using the age appropriate version of the Strengths and Difficulties Questionnaire (SDQ). The survey contains 6 questions asking about whether their behaviors are upsetting or distressing to the child. Parents rate as each question on a 4-point scale from not at all to a great deal. Scores are summed to yield a single score.
Parental acceptability the treatment | 12 months
  Parents will complete a survey asking them to rate the treatment program on 19 variables using a 7 point scale from negative to neutral to positive. Items will be summed to yield a program acceptability score

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Avellone, PhD, BCBA, LBA, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No